CLINICAL TRIAL: NCT03031054
Title: The Effect of Hyaluronic Acid in Patients With Carpal Tunnel Syndrome
Brief Title: The Effect of Hyaluronic Acid for Carpal Tunnel Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tri-Service General Hospital (Other)
Responsible Party: Principal Investigator, Yung-Tsan Wu, Attending Physician of Department of Physical Medicine and Rehabilitation, Tri-Service General Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HA for CTS
Record Dates: First submitted 2017-01-21; First posted 2017-01-25 (Estimated); Last update posted 2019-10-31 (Actual); Status verified 2019-10

CONDITIONS: Carpal Tunnel Syndrome
Keywords: Hydrodissection; hyaluronic acid
MeSH Terms: conditions — Carpal Tunnel Syndrome | interventions — Hyaluronic Acid; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- hyaluronic acid hydrodissection (Experimental): Ultrasound-guided hydrodissection with 2.5cc hyaluronic acid between carpal tunnel and median nerve.
  Interventions: Procedure: Sono-guided injection with hyaluronic acid
- Normal saline hydrodissection (Active Comparator): Ultrasound-guided hydrodissection with 2.5cc normal saline between carpal tunnel and median nerve.
  Interventions: Procedure: Sono-guided injection with normal saline

INTERVENTIONS:
Procedure: Sono-guided injection with hyaluronic acid — Sono-guided injection with hyaluronic acid (ARTZDispo, 25 mg/2.5 ml) between carpal tunnel and median nerve
  Arms: hyaluronic acid hydrodissection
Procedure: Sono-guided injection with normal saline — Sono-guided injection with 2.5cc Normal saline (0.9%) between carpal tunnel and median nerve
  Arms: Normal saline hydrodissection

SUMMARY:
Carpal tunnel syndrome (CTS) is the most common peripheral entrapment neuropathy with involving compression of the median nerve in the carpal tunnel. Rather than other progressive disease, CTS is characterized by remission and recurrence. The hydrodissection could decrease the entrapment of nerve to restore blood supply. In addition, the hyaluronic acid was proved to decrease adhension of soft tissue and nerve during operation. The investigators design a randomized, double-blind, controlled trial to assess the effect after ultrasound-guided hydrodissection with hyaluronic acid in patients with CTS.

DETAILED DESCRIPTION:
After obtaining written informed consent, patients with bilateral CTS will been randomized into intervention and control group. Participants in intervention group received one-dose ultrasound-guided hydrodissection with hyaluronic acid and control side received one-dose ultrasound-guided injection with normal saline. No additional treatment after injection through the study period. The primary outcome is Boston Carpal Tunnel Syndrome Questionnaire (BCTQ) and secondary outcomes include visual analog scale (VAS), cross-sectional area (CSA) of the median nerve, sensory nerve conduction velocity of the median nerve, and finger pinch strength. The evaluation was performed pretreatment as well as on the 2nd week, 1st, 3rd, 6th month and one year after the treatment.

ELIGIBILITY:
Inclusion Criteria:

* Age between 20-80 year-old.
* Diagnosis was confirmed using an electrophysiological study

Exclusion Criteria:

* Cancer
* Coagulopathy
* Pregnancy
* Inflammation status
* Cervical radiculopathy
* Polyneuropathy, brachial plexopathy
* Thoracic outlet syndrome
* Previously undergone wrist surgery or steroid injection for CTS

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2017-03-01 (Actual); Primary Completion 2019-10-28 (Actual); Study Completion 2019-10-28 (Actual)

PRIMARY OUTCOMES:
Change from baseline of severity of symptoms and functional status on 2nd week, 1st, 3rd, 6th month and one year after injection | Pre-treatment, 2nd week, 1st, 3rd, 6th month and one year
  Boston carpal tunnel syndrome questionnaire (BCTQ) is a frequently used patient-based questionnaire for measurement of CTS which encompasses two components. In total, 11 questions and 8 items were evaluated to rate the symptom severity scale (SSS) and functional status scale (FSS), respectively. Both subscales range from 1 to 5 with a higher score indicating a higher degree of disability. The mean of total SSS and FSS divided with each item score were used for further analysis.

SECONDARY OUTCOMES:
Change from baseline of pain on 2nd week, 1st, 3rd, 6th month and one year after injection | Pre-treatment, 2nd week, 1st, 3rd, 6th month and one year
  Digital pain severity or paresthesia/dysthesia was evaluated using visual analog scale (VAS). Pain score scale ranged from 0 to 10, with 10 indicating the most severe pain.
Change from baseline of cross-sectional area of the median nerve on 2nd week, 1st, 3rd, 6th month and one year after injection | Pre-treatment, 2nd week, 1st, 3rd, 6th month and one year
  Using the musculoskeletal sonogram to measure the cross-sectional area of the median nerve before treatment and multiple time frame after treatment.
Change from baseline of conduction velocity, amplitude of median nerve on 2nd week, 1st, 3rd, 6th month and one year after injection | Pre-treatment, 2nd week, 1st, 3rd, 6th month and one year
  electrophysiological study of the median nerve before treatment and multiple time frame after treatment.
Change from baseline of finger pinch on 2nd week, 1st, 3rd, 6th month and one year after injection | Pre-treatment, 2nd week, 1st, 3rd, 6th month and one year
  The finger pinch strength was measured using dynamometer (Fabrication Enterprises Inc., USA). The subject was seated with shoulder adducted and neutrally rotated with the elbow flexed at 90°. The forearm and wrist were positioned in a neutral position for the palmar pinch

CONTACTS AND LOCATIONS:
Overall Officials: Yung-Tsan Wu, MD, Principal Investigator — Department of Physical Medicine and Rehabilitation, Tri-Service General Hospital
Locations (2):
- Taiwan (2):
  - Department of Physical Medicine and Rehabilitation, Tri-Service General Hospital, Tai Chung Municipality, Neihu District
  - Department of Physical Medicine and Rehabilitation, Tri-Service General Hospital, Taipei, Neihu District

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Result] Ozgenel GY. Effects of hyaluronic acid on peripheral nerve scarring and regeneration in rats. Microsurgery. 2003;23(6):575-81. doi: 10.1002/micr.10209. PMID 14705074
- [Result] Burns JW, Skinner K, Colt J, Sheidlin A, Bronson R, Yaacobi Y, Goldberg EP. Prevention of tissue injury and postsurgical adhesions by precoating tissues with hyaluronic acid solutions. J Surg Res. 1995 Dec;59(6):644-52. doi: 10.1006/jsre.1995.1218. PMID 8538160
- [Result] Ozgenel GY, Filiz G. Effects of human amniotic fluid on peripheral nerve scarring and regeneration in rats. J Neurosurg. 2003 Feb;98(2):371-7. doi: 10.3171/jns.2003.98.2.0371. PMID 12593625
- [Result] Atzei A, Calcagni M, Breda B, Fasolo G, Pajardi G, Cugola L. Clinical evaluation of a hyaluronan-based gel following microsurgical reconstruction of peripheral nerves of the hand. Microsurgery. 2007;27(1):2-7. doi: 10.1002/micr.20299. PMID 17205576